CLINICAL TRIAL: NCT02065453
Title: Disposable Energy Sources and Operating Room Time for Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Mary Brigid Holloran-Schwartz, MD, Associate Professor, St. Louis University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22548
Record Dates: First submitted 2014-02-11; First posted 2014-02-19 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Benign Uterine Disease
Keywords: lap hysterectomy; Women in need of a lap hysterectomy for benign disease.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disposable Device - Left & Reusable Devices - Right (Other): One side of the uterine attachments would be transected using the disposable device (Ligasure, Covidien).
  Interventions: Device: disposable device (Ligasure, Covidien); Device: Reusable device
- Disposable Device - Right & Reusable Devices - Left (Other): One side of the uterine attachments would be transected using the reusable Robi bipolar and Storz laparoscopic
  Interventions: Device: disposable device (Ligasure, Covidien); Device: Reusable device

INTERVENTIONS:
Device: disposable device (Ligasure, Covidien) — One side of the uterine attachments would be transected using the disposable device (Ligasure, Covidien). . We will randomize the side for each energy source used on each side for every case. The number of "sides" performed by the attending surgeon will equal that of the less experienced resident surgeon.
  Other Names: disposable device (Ligasure made by Covidien).
Device: Reusable device — One side of the uterine attachments would be transected using the reusable Robi bipolar and Storz laparoscopic
  Other Names: Robi bipolar and Storz laparoscopic

SUMMARY:
Over 600,000 hysterectomies are performed each year nationwide. Over 99% of these are accomplished laparoscopically in the investigators current surgical practice to allow women a quicker recovery than a traditional large incision. Disposable laparoscopic devices have been developed to assist in the completion of hysterectomies. These disposable energy sources are only used once, but offer an improved safety and energy profile in that they reliably control bleeding with little damage to surrounding tissue and potentially save time. Reusable energy instruments can be sterilized and reused for multiple cases. Operating room time is expensive. The investigators calculate that if 6.7 minutes of time can be saved using the disposable device, Ligasure (Covidien), versus the reusable Robi bipolar and Storz Laparoscopic Shears, the time savings could justify the cost of the device.

DETAILED DESCRIPTION:
This will be a randomized, prospective study. The investigators study design would have each patient serve as their own control. One side of the uterine attachments would be transected using the disposable device, Ligasure (Covidien), and the other using the two reusable devices (Robi bipolar and Storz laparoscopic shears). It is the investigators standard practice that the attending surgeon is on the patient's left side while the resident physician is on the patients right. To eliminate the bias of surgical experience, the investigators will randomize the energy source used on each side for every case. Therefore, the number of cases performed by the attending surgeon with the disposable or reusable energy sources, will equal that of the less experienced resident surgeon.

The primary endpoint of this study would be the time difference between cauterizing one side of the uterine attachments, from the round ligament to the uterine artery on one side, to the time detaching the same tissues on the other side. The vesico-uterine peritoneum or "bladder flap", will always be transected from the left for consistency. Sealed, opaque envelopes will be randomized to determine which side of the uterus will get the single disposable instrument, and which will get the 2 reusable instruments.

A time savings of 6.7 minutes for the total case can also be explained by a 3.35 minute time savings PER SIDE of the uterine attachments, given each uterus has two "sides". There is no pre-existing data on time needed for coagulation and cutting of the vascular tissues. Based on experience, the investigators estimate that it takes on average about 20 min total time for vessel sealing, with an estimated variability that approximately 70% of the time, vessel sealing is done within 35 minutes. Given these estimates, and using a power of 0.8, the sample size needed is 45.

The primary endpoint of surgical time will be initially assessed for each individual patient by determining the difference between the half of the laparoscopic hysterectomy procedure performed with the disposable device, specifically the Ligasure (Covidien) and the half of the laparoscopic hysterectomy procedure performed with the two reusable devices (Robi Bipolar and Storz laparoscopic shears) and determining if the mean difference score summed across all patients differs significantly from zero. Subsequent analyses will examine surgical times for attending physicians and residents separately where those using the disposable device are compared to those using the two reusable devices with independent students t test or the Kolmogorov-Smirnov test depending on the normality of the distributions. Parallel analyses will be performed for the secondary endpoint of estimated blood loss. Secondary endpoints of organ damage and other categorical intraoperative complications will be compared between the disposable and reusable device groups using chi-square and Fisher's Exact test.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years of age
* Scheduled for laparoscopic hysterectomy (prospectively)

Exclusion Criteria:

* Under 21 years of age
* Known or anticipated malignancy

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Holloran-Schwartz, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

RESULTS

PARTICIPANT FLOW:
Groups:
- Disposable Device - Left & Reusable Devices - Right: 27 women were randomized to attending physicians using the disposable device on the left and reusable devices on the right.
- Disposable Device - Right & Reusable Devices - Left: 25 women were randomized to attending physicians using the disposable device on the right and reusable devices on the left
Period: Overall Study
Arm/Group | Disposable Device - Left & Reusable Devices - Right | Disposable Device - Right & Reusable Devices - Left
Started | 27 | 25
Completed | 24 | 21
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Disposable Device Left and Resusable Devices Right: 27 women were randomized to receive disposable device left and resusable devices right
- Disposable Device Right and Reusable Devices Left: 25 women were randomized to receive disposable device right and reusable devices left
- Total: Total of all reporting groups
Arm/Group | Disposable Device Left and Resusable Devices Right | Disposable Device Right and Reusable Devices Left | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [24 to 48] | 39 [24 to 48] | 39 [24 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study is Time Difference Between Cauterizing One Side of the Uterine Attachments, From the Round Ligament to the Uterine Artery on One Side, to the Time Detaching the Same Tissues on the Other Side
Description: duration of surgery
Time Frame: Primary outcome study data is collected with the first incision and completed with skin closure at the completion of the surgery.
Population: Uterine Vessel Desiccation and Electrosurgical Cutting Time (min)
Measure: Median (Full Range); unit: minutes
Groups:
- Disposable; Reusable: Uterine Vessel Desiccation and Electrosurgical Cutting Time (min) Resident and Attending Physicians Combined
Arm/Group | Disposable | Reusable
Number analyzed (Participants) | 45 | 45
minutes | 8.4 [8.4 to 8.7] | 14.6 [12.5 to 16.7]
Statistical Analysis 1: Comparison: Disposable vs Reusable; The data will be analyzed using linear regression, Kolmogorov-Smirnov test, and chi-square analysis; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 weeks post op, surgical procedure
Description: No adverse events were noted
Groups:
- Disposable or Reusable Energy Sources: Each patient serve as their own control. One side of the uterine attachments would be transected using the disposable device, the Ligasure, and the other using the two reusable devices, the Robi bipolar and Storz laparoscopic shears. It is our standard practice that the attending surgeon is on the patient's left side while the resident physician is on the patients right. To eliminate the bias of surgical experience, we will randomize the energy source used on each side for every case. Therefore, the number of cases performed by the attending surgeon with the disposable or reusable energy sources, will equal that of the less experienced resident surgeon.
Arm/Group | Disposable or Reusable Energy Sources
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No